CLINICAL TRIAL: NCT05004207
Title: Oro-cecal Transit Time in Healthy Indian Subjects Using Scintigraphy and Its Correlation With Lactulose Hydrogen Breath Test- A Pilot Study
Brief Title: Study of Oro-cecal Transit Time in Healthy Subjects Using Scintigraphy and Lactulose Hydrogen Breath Test.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, Senior Consultant, Asian Institute of Gastroenterology, India
Other Study IDs: AIG/IEC-BH&R 15/06.2021-02
Record Dates: First submitted 2021-08-04; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Small Bowel Disease; Motility Disorder; Irritable Bowel Syndrome
Keywords: Small bowel disease; Orocaecal transit time; nuclear scintigraphy; lactulose hydrogen breath test
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 99mTc Scintigraphy — After fasting for at least 8 to 12 hours, standardized meal mixed with 99mTc-sulfur colloid radiolabeled test will be administered as quickly as possible, optimally within 10 min. Imaging will be obtained with Siemens SYMBIA E dual head (SPECT) scanner in a format of at least 128 x 128 pixels. Anterior and posterior planar images (or a single left anterior oblique image) with the distal esophagus, stomach, and proximal small bowel in the field of view will be obtained for 1 min immediately after ingestion of the test meal and repeated images will be obtained in the same projections with 2 min static images at hourly intervals up to 6 h and at 24 hours as was used for the initial images.
  Next day LHBT will be performed after at least 12 hours of fasting. Following administration of test substrate (Lactulose 10 grams) with one cup of water, breath samples will be analyzed for hydrogen every 15 minutes for 1 hour followed by every half hour for next 2 hour with LACTOFEN 2 device.
  Other Names: Lactulose Hydrogen Breath test

SUMMARY:
Radionuclide scintigraphy is the gold standard technique to interpret OCTT but there is no normative data available for its interpretation in Indian population. Previous studies to determine OCTT have all been done with LHBT, which has many limitations. Besides there are few small comparative studies between scintigraphy and LHBT, that too not in Indian population. The aim of this study is to validate LHBT to measure OCTT compared with scintigraphy and to standardize the normal OCTT in healthy individuals

DETAILED DESCRIPTION:
1. INTRODUCTION Oro-caecal transit time (OCTT) can be defined as time taken for the meal to reach from oral cavity to caecum and how long it takes for food to pass through small intestines. It's important because it influences how efficiently nutrients are absorbed from food and influences fermentation associated with healthy gut flora. Short transit time may be due to inflammation caused by intestinal infection, food allergies, or by absence of healthy intestinal flora. Long transit time is usually due to eating too much refined and processed foods, low thyroid, dehydration, lack of dietary fibre, serotonin deficiency and insufficient salt intake Several factors affect the oro-caecal transit time such as: physiological (age, sex, menstrual cycle), usage of stimulants (coffee, alcohol, cigarette smoking), as well as pathological conditions. Patients can have gastrointestinal symptoms, which may be secondary to small intestinal dysmotility which can be achieved by interpretation of oro- caecal transit time. Thus measurement of OCTT helps in various GI diseases eg. chronic constipation, chronic diarrhoea, Dyspepsia, Irritable bowel syndrome, chronic idiopathic intestinal pseudo-obstruction or functional recto-sigmoid obstruction, scleroderma, celiac disease & Malabsorption syndrome. Two techniques are available to assess oro-cecal transit time, Lactulose hydrogen breath test and Radionuclide scintigraphy, where latter is the gold standard technique to interpret OCTT.
2. RATIONALE Radionuclide scintigraphy is the gold standard technique to interpret OCTT but there is no normative data available for interpretation of OCTT in Indian population. Previous studies to determine OCTT have all been done with LHBT, which has many limitations. Besides there are few small comparative studies between scintigraphy and LHBT, that too not in Indian population. Interpretation of OCTT helps in assessment of various GI disorders which may be secondary to small intestinal dysmotility having gastrointestinal symptoms.
3. STUDY POPULATION- 50 healthy asymptomatic subjects
4. DESIGN AND DURATION OF THE STUDY- It will be a pilot study. The study duration will be till completion of data collection for 50 subjects.
5. METHODOLOGY- 5a. SUBJECT RECRUITMENT - Healthy volunteers

5b. RANDOMIZATION AND BLINDING- N/A

5c. STUDY METHODS- This observational study will be conducted among 50 patients of both sexes after obtaining ethical clearance from institutional human ethical committee. Study participants will be of the age more than 18 years. Exclusion criteria will consist of thoracic or digestive foregut surgery, alcohol consumption >40 g/day, use of medications that alter intragastric acidity or esophageal motility, as well as history of diabetes mellitus, thyroid disorder, neurological disorders or other chronic gastrointestinal disease.

5d. STUDY PROCEDURE- Subjects will be advised to stop any medications that affect GI motility 2 days prior to testing and avoid strenuous exercise and cigarette smoking on the day of test. After fasting for at least 8 to 12 hours, standardised meal - 3 idli plus curd mixed with 18.5-37 Minimum Base Quantity (MBq) (0.5-1 mCi) of 99mTc-sulfur colloid radiolabelled test meal will be administered as quickly as possible, optimally within 10 min. Imaging will be obtained with Siemens Symbia E dual head scanner in a format of at least 128 x 128 pixels using a general-purpose collimator or a low energy high-resolution collimator The photopeak settings are 20% at the 140-keV (kiloelectron volt) peak for 99mTc. Anterior and posterior planar images (or a single left anterior oblique image) with the distal oesophagus, stomach, and proximal small bowel in the field of view will be obtained for 1 min immediately after ingestion of the test meal and Repeated images will be obtained in the same projections with 2 min static images at hourly intervals up to 6 h and 24 h, as was used for the initial images.

Next day after at least 12 hours of fasting with no strenuous exercise and cigarette smoking on the day of test, with no antibiotics 4 weeks prior to testing and no prokinetic drug or laxatives 2 weeks prior to testing. Following administration of test substrate (Lactulose 10 grams) with one cup of water, breath samples will be analysed for hydrogen every 15 minutes for 1 hour followed by every ½ hour for next 2 hour with LACTOFEN 2 device.

5e. METHODS OF ASSESSMENT-.The analysis process will consist of:

1. Interpretation of oro-caecal transit time with scintigraphy i.e by the percentage accumulation of 99mTc in the caecum
2. Interpretation of oro-caecal transit time with LHBT i.e the time interval between ingestion of lactulose and rise in breath hydrogen 20 ppm above basal
3. Co-relation of oro-caecal time between scintigraphy and LHBT

   6. Sample Size Calculaion- It will be a pilot study. The study duration will be till completion of data collection for 50 subjects.

   7. Statistical Analysis- Data will be expressed as median and percentile values (5th, 25th, 75th and 95th percentiles). Depending on normality of distribution, we will use either paired Student's t-test or Mann-Whitney U test for paired comparison. Likewise, we will use one way analysis of variance with Tukey test or Kruskal-Wallis, followed by Dunn's test as appropriate. Upper limit of normal will be defined as the 95th percentile of normal values. P≤0.05 will be considered statistically significant.

   8. ETHICAL JUSTIFICATION OF THE STUDY - Both the procedure being done in this study are considered safe and not associated with any major adverse event. But there is very minimal risk of radiation exposure in radionuclide scintigraphy study, which is less than exposure to a chest X ray.There is no normative data available for interpretation of OCTT in Indian subjects using nuclear scintigraphy. The commonly used test for measurement of OCTT, i.e LHBT has also not been validated in Indian subjects as compared to the scintigraphy. This study will help us give a reference value for OCTT, which could be used for defining altered small bowel transit time.

ELIGIBILITY:
Inclusion Criteria:

• Healthy individual > 18 years of age with no comorbidities

Exclusion Criteria:

* Thoracic or digestive foregut surgery,
* Alcohol consumption >40 g/day,
* Use of medications that alter intragastric acidity or oesophageal motility
* History of diabetes mellitus, thyroid disorder
* Neurological disorders
* Chronic gastrointestinal disease
* Any subject with upper GI symptoms like pain, burning, belching, bloating, dysphagia & aerophagia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individual > 18 years of age with no comorbidities
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Oro-caecal transit time (OCTT) using lactulose hydrogen breath test (LHBT) and scintigraphy study. | six months
  LHBT is the commonly used test for OCTT, but it has fallacies, since it itself increase intestinal motility, so this study aims to validate LHBT with scintigraphy which is the gold standard test.

SECONDARY OUTCOMES:
Normative data for OCTT using nuclear scintigraphy in healthy indian population. | six months
  There is no reference values for nuclear scintigraphy in healthy indian patients. The study will help generate data to give reference values for OCTT using scintigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh kalapala, MBBS, MD, DM, Study Director — Senior Consultant; Pratik Chhabra, MBBS, MD, Principal Investigator — Fellow; Suneetha B, MBBS, MD, DM, Principal Investigator — Consultant
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Result] Miller MA, Parkman HP, Urbain JL, Brown KL, Donahue DJ, Knight LC, Maurer AH, Fisher RS. Comparison of scintigraphy and lactulose breath hydrogen test for assessment of orocecal transit: lactulose accelerates small bowel transit. Dig Dis Sci. 1997 Jan;42(1):10-8. doi: 10.1023/a:1018864400566. PMID 9009110
- [Result] Yu D, Cheeseman F, Vanner S. Combined oro-caecal scintigraphy and lactulose hydrogen breath testing demonstrate that breath testing detects oro-caecal transit, not small intestinal bacterial overgrowth in patients with IBS. Gut. 2011 Mar;60(3):334-40. doi: 10.1136/gut.2009.205476. Epub 2010 Nov 26. PMID 21112950
- [Result] Ning Y, Lou C, Huang Z, Chen D, Huang H, Chen L, Zhang B, Dai N, Zhao J, Zhen X. Clinical value of radionuclide small intestine transit time measurement combined with lactulose hydrogen breath test for the diagnosis of bacterial overgrowth in irritable bowel syndrome. Hell J Nucl Med. 2016 May-Aug;19(2):124-9. doi: 10.1967/s002449910365. Epub 2016 Jun 22. PMID 27331205
- [Result] Zhao J, Zheng X, Chu H, Zhao J, Cong Y, Fried M, Fox M, Dai N. A study of the methodological and clinical validity of the combined lactulose hydrogen breath test with scintigraphic oro-cecal transit test for diagnosing small intestinal bacterial overgrowth in IBS patients. Neurogastroenterol Motil. 2014 Jun;26(6):794-802. doi: 10.1111/nmo.12331. Epub 2014 Mar 18. PMID 24641100
- [Result] Gilmore IT. Orocaecal transit time in health and disease. Gut. 1990 Mar;31(3):250-1. doi: 10.1136/gut.31.3.250. No abstract available. PMID 2182399